CLINICAL TRIAL: NCT04256603
Title: Evaluation of Initiation Time on the Efficacy of Gabapentin in Treating Neuropathic Pain in Spinal Cord Injury (SCI)
Brief Title: Evaluation of Initiation Time on the Efficacy of Gabapentin in Treating Neuropathic Pain in SCI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Chong Kim, PI, MetroHealth Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB19-00117
Record Dates: First submitted 2020-02-01; First posted 2020-02-05 (Actual); Results first posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Spinal Cord Injuries; Neuropathic Pain
Keywords: neuropathic pain; spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia | interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Gabapentin early (Other): Gabapentin prior to admission
  Interventions: Drug: Gabapentin
- Gabapentin late (Other): Gabapentin during admission
  Interventions: Drug: Gabapentin
- No gabapentin (Other): No gabapentin
  Interventions: Other: No gabapentin

INTERVENTIONS:
Drug: Gabapentin — Timing of gabapentin initiation
  Arms: Gabapentin early; Gabapentin late
Other: No gabapentin — No gabapentin
  Arms: No gabapentin

SUMMARY:
Neuropathic pain is a common complaint in those with spinal cord injury (SCI) that has a significant negative effect on quality of life. Efficacy of various treatments, however, remains controversial. There is evidence to support that gabapentin and pregabalin have some benefit in reducing neuropathic pain. Gabapentin is effective in the management of symptoms and concerns related to SCI including motor recovery, spasticity, and mood among others. This makes gabapentin an important pharmacologic intervention, which compels providers to define treatment guidelines related to its use. One aspect of which should relate to the timing of initiation of therapy. The goal of this study is to determine whether timing of initiation of treatment with gabapentin will decrease prevalence and intensity of neuropathic pain.

DETAILED DESCRIPTION:
Neuropathic pain is a common complaint in those with spinal cord injury (SCI) that has a significant negative effect on quality of life. This makes the treatment of neuropathic pain a priority in the SCI population. Efficacy of various treatments, however, remains controversial. There is evidence to support that gabapentin and pregabalin have some benefit in reducing neuropathic pain. Other positive effects of gabapentin on those with SCI have also been demonstrated. However, there has not been a study on the influence of timing of initiation of gabapentin on the efficacy of using it to treat neuropathic pain in the SCI population. Such a finding could change the standard of care in treatment of acute SCI.

The pooled prevalence of neuropathic pain post spinal cord injury is 53%. Not only common, neuropathic pain is pervasive, affecting aspects of patients' lives including sleep, physical function, and mood that in turn impact their activities- work and recreational alike. Thus, neuropathic pain management contributes to quality of life for a majority of people with SCI.

Although a high priority, the treatment of neuropathic pain in SCI remains notoriously difficult. Treatments options may be divided into pharmacologic and non-pharmacologic. Pharmacologic agents studied include amitriptyline, gabapentin, pregabalin, opiates, lidocaine, ketamine, valproate, lamotrigine, levetiracetam and carbamazepine; the most studied of which are amitriptyline, gabapentin, and pregabalin.

Gabapentin's potential is not limited to neuropathic pain management, making it a particularly compelling treatment option in the population with acute SCI. Gabapentin leads to improvement in total motor scores, reduced spasticity, reduced autonomic dysreflexia, and improved mood. Animal models suggest it may be neuroprotective in the acute phase of injury. In those who undergo spine surgery, regardless of presence of SCI, gabapentin given perioperatively leads to reduced opiate use and decreased pain in post-operative period. Additionally, when compared to narcotic alternatives, gabapentin has minimal side effects.

Neuropathic pain in SCI is common, impactful, and difficult to treat. Gabapentin is effective in the management of symptoms and concerns related to SCI including motor recovery, spasticity, and mood among others. This makes gabapentin an important pharmacologic intervention, which compels providers to define treatment guidelines related to its use. One aspect of which should relate to the timing of initiation of therapy. The goal of this study is to determine whether early initiation of treatment with gabapentin will decrease average pain scores and opiate use when comparted to late initiation of treatment with gabapentin in the population with acute SCI. Gabapentin, although used commonly, is not started in all patients with acute SCI but is often started at the onset of neuropathic pain. If gabapentin is found to be more effective when initiated early, it would be reasonable to start gabapentin immediately following acute SCI in all patients in whom it is not otherwise contraindicated.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of acute spinal cord injury
2. Admission to acute inpatient rehabilitation

Exclusion Criteria:

1. Unable to communicate verbally or by writing, unable to follow basic instructions, or unable to answer questions regarding their symptoms

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C Kim, Principal Investigator — Metro Health, Michigan
Locations (1):
- MetroHealth, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Gabapentin Group: The arm included subjects who met all inclusion criteria, those with acute spinal cord injury admitted to acute care hospital and were approved and admitted to inpatient rehabilitation unit. All subjects in this group were started on Gabapentin prior to admission and continued during care. All subjects were screened with questionnaires with data collection based on electronic medical records.
- No Gabapentin Group: The arm included subjects who met all inclusion criteria, those with acute spinal cord injury admitted to acute care hospital and were approved and admitted to inpatient rehabilitation unit. All subjects in this group were started on Gabapentin during inpatient rehabilitation admission and continued during care. All subjects were screened with questionnaires with data collection based on electronic medical records. g care.
Period: Overall Study
Arm/Group | Gabapentin Group | No Gabapentin Group
Started | 21 | 6
Completed | 21 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Gabapentin: Gabapentin prior to admission
  Gabapentin: Timing of gabapentin initiation
- No Gabapentin: Gabapentin during admission
  Gabapentin: Timing of gabapentin initiation
- Total: Total of all reporting groups
Arm/Group | Gabapentin | No Gabapentin | Total
Number analyzed (Participants) | 21 | 6 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 6 | 27
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 16 | 5 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 6 | 27
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Neuropathic Pain
Description: To determine if the time from injury influences the prevalence of neuropathic pain in acute SCI. Average of the pain during the previous 7 days on self-identified nerve or neuropathic pain levels (0-10) on 5 different measurements at the time of discharge on the Neuropathic Pain Scale. 0 being best (no pain)- 10 being worst pain. Total score range from 0 to 50.
Time Frame: Through completion of the study, up to 4 weeks after injury.
Population: 21 subjects were enrolled in the group treated with gabapentin, vs 6 in then no gabapentin
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin Group | No Gabapentin Group
Number analyzed (Participants) | 21 | 6
units on a scale | 13.3 (18.8) | 15.6 (18.0)
Statistical Analysis 1: Comparison: Gabapentin Group vs No Gabapentin Group; wilcox two sample test; Test type: Other; p = 0.67, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 9 months
Description: during hospital stay until discharge
Arm/Group | Gabapentin Group | No Gabapentin Group
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/6
Other Adverse Events (participants affected / at risk) | 0/21 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/03/NCT04256603/Prot_SAP_ICF_002.pdf